CLINICAL TRIAL: NCT02646540
Title: AiDing Diuresis wIth Tolvaptan (ADD-IT)
Acronym: ADD-IT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Divya Gupta, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00080051
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Cardiomyopathy; Congestive Heart Failure
MeSH Terms: conditions — Cardiomyopathies; Heart Failure | interventions — Tolvaptan; Diuretics; Furosemide; Metolazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tolvaptan 30 mg and IV Lasix (Experimental): Participants admitted to the hospital and diagnosed with acutely decompensated heart failure (ADHF) will receive 30 mg of tolvaptan concomitantly with their standard dose of diuretics.
  Interventions: Drug: Tolvaptan 30 mg + IV Diuretics
- Metolazone 5mg and IV Lasix (Active Comparator): Participants admitted to the hospital and diagnosed with acutely decompensated heart failure (ADHF) will receive 5mg metolazone concomitantly with their standard dose of diuretics.
  Interventions: Drug: Metolazone 5 mg + IV Diuretics
- IV Lasix (Active Comparator): Participants admitted to the hospital and diagnosed with acutely decompensated heart failure (ADHF) will receive two and a half (2.5) times their standard dose of diuretics.
  Interventions: Drug: 2.5 times the Diuretics Dose

INTERVENTIONS:
Drug: Tolvaptan 30 mg + IV Diuretics — Participants will receive oral daily tolvaptan 30 mg concomitantly with their standard dose of intravenous (IV) diuretics for the duration of their hospitalization.
  Other Names: Tolvaptan (Samsca) and Lasix (Furosemide)
  Arms: Tolvaptan 30 mg and IV Lasix
Drug: Metolazone 5 mg + IV Diuretics — Participants will receive oral daily metolazone 5 mg concomitantly with their standard dose of intravenous (IV) diuretics for the duration of their hospitalization.
  Other Names: Metolazone (Zaroxolyn) and Lasix (Furosemide)
  Arms: Metolazone 5mg and IV Lasix
Drug: 2.5 times the Diuretics Dose — Participants will receive two and a half (2.5) times their standard dose of intravenous (IV) diuretics for the duration of their hospitalization.
  Other Names: Lasix (Furosemide)
  Arms: IV Lasix

SUMMARY:
The purpose of this study is to test the use of tolvaptan (commercial name Samsca) when given in addition to intravenous (IV) diuretics early during an episode of acute heart failure. It will be compared to a high dose of IV diuretics alone or the use of metolazone in addition to IV diuretics. The investigators are looking to see if there is improvement in the symptoms and outcomes of persons with acute heart failure.

DETAILED DESCRIPTION:
This is a single-center, randomized trial to assess the effects of 30 mg daily of tolvaptan when given concomitantly with home dose of diuretic (Lasix equivalent) intravenously (IV) versus 5mg daily of metolazone given concomitantly with home dose of diuretic (Lasix equivalent) IV, versus 2.5 times home dose of diuretic (Lasix equivalent) IV in participants hospitalized for acutely decompensated heart failure (ADHF).

ELIGIBILITY:
Inclusion Criteria:

* Participants hospitalized for worsening acute heart failure and randomized within 36 hours of initial presentation
* New York Heart Association (NYHA) Class III or IV on admission to the hospital with at least 1 month history of treated heart failure
* Able to understand content of and willing to provide written informed consent

The participant must have signs of extracellular volume expansion, defined as two or more of the following four signs or symptoms:

* signs of RHF (right heart failure) (jugular venous distention, pitting edema, or (≥1+), ascites and/or signs of LHF (left heart failure) (pulmonary congestion on chest x-ray, pulmonary rales)
* Brain Natriuretic Peptide (BNP) > 450
* serum sodium < 140 mEq/L

Exclusion Criteria:

* Positive urine pregnancy test for women of child bearing potential
* Inability to provide written informed consent
* Cardiac surgery within 60 days prior to study randomization
* Acute Coronary Syndrome (ACS) or percutaneous coronary intervention within 30 days prior to study randomization
* Planned revascularization procedures, cardiac mechanical support implantation, cardiac transplantation, or other cardiac surgery within 30 days following study randomization
* Planned electrophysiologic (EP) device implantation within 7 days following study randomization
* Subjects who are on cardiac mechanical support
* Co- morbid condition with an expected survival less than six months
* History of a cerebrovascular accident within the last 30 days
* Hemodynamically significant uncorrected primary cardiac valvular disease
* Hypertrophic cardiomyopathy (obstructive or non-obstructive)
* Uncorrected thyroid disease, active myocarditis or known amyloid cardiomyopathy
* History of primary significant liver disease or acute hepatic failure, defined as 3x upper limit of normal (ULN)
* Chronic uncontrolled diabetes mellitus with Hemoglobin A1C > 10%
* Supine systolic arterial blood pressure < 90 mmHg
* Serum creatinine > 3.5 mg/dL or undergoing dialysis
* Hemoglobin < 9 g/dL
* History of hypersensitivity and/or idiosyncratic reaction to benzazepine derivatives (such as benazepril)
* Inability to take oral medications
* Participation in another clinical drug or device trial where the last dose of drug was within the past 30 days or an investigational medical device is currently implanted
* Previous exposure to tolvaptan within 7 days prior to randomization
* Subjects with refractory, end-stage, heart failure defined as subjects who are appropriate candidates for specialized treatment strategies, such as ventricular assist devices, continuous positive IV inotropic therapy, or hospice care
* Ultrafiltration within 7 days prior to randomization or planned.
* Active gout

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Length of Hospitalization Measured in Days | Duration of Hospitalization (Average of Five Days)
  The number of days hospitalized until discharge.

SECONDARY OUTCOMES:
Change in Body Weight | Baseline (hospital admission), Discharge (Average of 5 Days)
  The difference in body weight from hospital admission to discharge measured in kilograms.
Total Diuretic Dose | Up to Five Days
  The total dose of diuretics given throughout the duration of hospitalization measured in milligrams (mg).
Change in estimated glomerular filtration rate (eGFR) | Baseline (hospital admission), Discharge (Average of 5 days)
  The difference in eGFR from baseline (hospital admission) to discharge.
Number of Days Alive | Post Hospital Discharge (30 days)
  The number of days participants remain alive over thirty days after hospital discharge.
Rate of Re-Hospitalization | 30 Days Post Hospitalization
  The number of participants re-hospitalized for worsening heart failure or death at 30 days.
Number of Electrolyte Imbalance Related Adverse Events | Duration of Hospitalization (Average of Five Days)
  The number of adverse events due to electrolyte imbalance throughout the duration of hospitalization.
Number of Participants Requiring Electrolyte Repletion | Duration of Hospitalization (Average of Five Days)
  The number of participants that require electrolyte repletion throughout the duration of hospitalization.
Change in Sodium Level | Baseline (hospital admission), Discharge (Average of 5 days)
  The difference in sodium levels from baseline to hospital discharge measured in milliequivalents per liter (mEqL).

CONTACTS AND LOCATIONS:
Overall Officials: Divya Gupta, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia